CLINICAL TRIAL: NCT05284240
Title: Prospective, Multi-center, Single-arm Study of the Auryon Laser System for Treatment of Below-the-Knee (BTK) Arteries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Cardiovascular Research Foundation (Other)
Collaborators: Angiodynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCRF-P003-2021
Record Dates: First submitted 2022-02-02; First posted 2022-03-17 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, single arm study Patients with symptomatic peripheral vascular disease who underwent infrapopliteal percutaneous intervention using the Auryon laser system 4 sites in United States
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Auryon Laser Treatment Arm (Experimental): Auryon Laser to be used on target lesion in the below the knee artery.
  Interventions: Device: Auryon Laser System

INTERVENTIONS:
Device: Auryon Laser System — The Auryon BTK Study is a prospective, single arm multicenter study evaluating the safety and procedural effectiveness of the Auryon laser in treating infrapopliteal disease in patients with critical limb ischemia and claudication.
  The primary exposure of interest for this study is the use of the AURYON system for atherectomy.

SUMMARY:
The Auryon Laser Atherectomy System has been cleared by the FDA to treat infrainguinal arterial disease including in-stent restenosis

DETAILED DESCRIPTION:
To observe the treatment effects of the Auryon Laser Atherectomy System in treating Infrapopliteal peripheral arterial disease

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years of age or older. 2. Critical limb ischemia (CLI) in the target limb from the distal segment (P3) of the popliteal artery to the ankle joint prior to the study procedure with Rutherford Category 4-5 in the target limb from the distal segment (P3) of the popliteal artery to the ankle joint prior to the study procedure.

3. Patient has signed approved informed consent. 4. Patient is willing to comply with the follow-up evaluations Angiographic Inclusion Criteria

1. Target lesions(s) must be viewed angiographically and have ≥50% stenosis. More than one lesion can be included in the same vessel.
2. Only 1 target vessel is included in the study.
3. Intraluminal crossing of the lesion. If this is not certain, IVUS may be used to verify this per operator's discretion.

Target Lesion reference vessel diameter (RVD) between 1.5 mm - 4.5 mm. by investigator estimate.

4. Target lesion is denovo or restenotic.

-

Exclusion Criteria:

1. Target lesion is in a vessel graft or synthetic graft.
2. Subjects requiring dialysis.
3. Subject is unable to understand the study or has a history of non-compliance with medical advice.
4. Subject is unwilling or unable to sign the Informed Consent Form (ICF)
5. Subject is currently enrolled in another clinical investigational study that might clinically interfere with the current study endpoints.
6. Subject has a known sensitivity to contrast media and the sensitivity cannot be adequately pre-medicated for.
7. Subject has a CVA or TIA within 4 weeks prior to the Auryon procedure.
8. Planned Use of another debulking device or specialty balloons before or after the Auryon laser during the index procedure
9. Patient has any planned surgical intervention or endovascular procedure ≤14 days after the index procedure or had these procedures in the past 14 days
10. Life expectancy of less than one year judged by the investigator
11. Patient unable to take anticoagulant or antiplatelet agents
12. Platelet count less than 80,000K or bleeding disorders
13. Subject is suspected of having an active systemic infection.
14. Patient enrolled once already in the protocol
15. Planned major amputation of either leg.
16. Acute limb ischemia
17. Current Covid-19 Infection or history of Covid-19 in the past 30 days.
18. Subject is pregnant or planning on becoming pregnant.
19. Vulnerable patients who are unable to give informed consent on their own Pregnant and Vulnerable Populations. There will be no female patients who are pregnant or any vulnerable populations enrolled in the study.
20. Subject experiencing ongoing cardiac problems that per the investigator judgment would not make the subject ideal per the procedure
21. Subject has evidence of intracranial or gastrointestinal bleeding within the past 3 Angiographic Exclusion Criteria

1. Failure to treat clinically significant inflow lesions in the contralateral iliac, ipsilateral iliac, femoral, or P1-P2 segments of the popliteal arteries with ≤ 30 % residual stenosis, and no serious angiographic complications (e.g., embolism) 2. Failure to successfully treat significant non-target infra-popliteal lesions prior to treatment of the target lesion. Successful treatment is defined as obtaining ≤ 50 % residual stenosis with no serious angiographic complications (e.g., embolism).

3. Failure to successfully cross the guidewire across the target lesion; successful crossing is defined as tip of the guidewire distal to the target lesion in the absence of flow limiting dissections or perforations.

4. In-stent restenosis.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
The Primary Safety Endpoint: | 30 days
  Major Adverse Limb Events (MALE) + Post-Operative Death (POD) at 30 days, as adjudicated by the CEC, defined as a composite of:
  1. All-cause death
  2. Above-ankle amputation of the index limb
  3. Major reintervention (new bypass graft, jump/interposition graft revision, or thrombectomy/thrombolysis) of the index limb involving a BTK artery
The Primary Performance Endpoint: | Index Procedure
  Procedure Success defined as ≤30% residual stenosis for the treated segment of the vessel without serious angiographic complications (flow-limiting dissection (D to F), perforation, distal embolization, or acute vessel closure after final treatment, as assessed by the angiographic core lab.

SECONDARY OUTCOMES:
Serious angiographic complications | Index Procedure
  flow-limiting dissection (D to F, perforation, distal embolization, or acute vessel closure) as assessed by the angiographic core lab
Technical success | Index Procedure
  defined as residual stenosis ≤50% in the target lesion after Auryon laser and prior to adjunctive balloon treatment without significant angiographic complications, as assessed by the angiographic core lab
Primary patency at 6 and 12 month | 6 and 12 months
  s defined as the absence of both total occlusion (100% diameter stenosis by DUS) in all of the target lesions, as well as a Clinically-Driven Target Lesion Revascularization (CD-TLR) (definition in D below). An alternative patency analysis will be done with patency defined as the presence of significant restenosis at the treated site using PSVR of ≤ 2.4 as the threshold for patency and absence of CD-TLR
Clinically Relevant Target Lesion Revascularization | 12 months
  (CD-TLR) at 30 days, 3, 6, and 12 months defined as recurrence of symptoms (worsening by one Rutherford Becker Category from post index procedure) with an objective evidence of obstructive disease (occlusion or PSVR > 2.4 by DUS; or ABI change by 0.15 from post procedure ABI)
Major Adverse Events (MAE) | 30 days
  Composite
  * Need for emergency surgical revascularization of target limb
  * Unplanned target limb major amputation (above the ankle)
  * Symptomatic thrombus or distal emboli that require surgical, mechanical, or pharmacologic means to improve flow, and extend hospitalization
Perforations | Index Procedure
  Perforations that require an intervention
Walking impairment questionnaire | 30 days, 3, 6, and 12 months
  reported as change from baseline
EQ-5D-5L Questionnaire | 30 days, 3, 6, and 12 months
  reported as change from baseline
Ankle-brachial Index (ABI) or Toe-brachial Index (TBI) | 30 days, 6 and 12 months
  reported as change from baseline
Rutherford Category | 30 days, 3, 6, and 12 months
  reported as change from baseline
Subgroup analysis stratified by IVUS | Index Procedure
  Subgroup analysis stratified by IVUS vs non IVUS patients for the primary performance endpoint and the following secondary endpoints: Final Balloon Size used to dilate lesion post laser, CD-target lesion revascularization and clinical patency
Healed Wounds | 30 days, 3, 6, and 12 months
  Number of healed wounds
Mean Lesion Diameter | Index Procedure
  IVUS subgroup: 20 patients. All will be evaluated for MLA pre and post laser and post final treatment.
Total Dissections | Index Procedure
  The presence and number of dissections will be classified based on iDissection classification

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Shammas, Principal Investigator — Midwest Cardiovascular Research Foundation
Locations (2):
- United States (2):
  - Palm Vascular Centers, Miami Beach, Florida
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa

IPD SHARING:
Plan to Share IPD: No